CLINICAL TRIAL: NCT02859805
Title: Validation of a Diagnostic Self-assessment Scale Non-motor Fluctuations at the Parkinson's Patient
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_3341 - 1726
Record Dates: First submitted 2016-07-28; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: validation of a diagnostic tool severity of non-motor symptoms in Parkinson patients

SUMMARY:
The objective of this study is to validate a diagnostic tool severity of these common non-motor manifestations, disturbing and little recognized as a self-questionnaire. This assessment tool used on different subgroups of patients (free from any treatment at an early stage of the disease and the stage of motor complications) will better understand the natural history of the non-motor fluctuations (FNM)

ELIGIBILITY:
Inclusion Criteria:

Patient aged 30 or over Patient having an Parkinson's disease Patient hospitalized in one of the clinical sites participating in the project Patient have agreed to participate in the study subject that masters the French language and able to fulfill the self-questionnaire.

Exclusion Criteria:

Patient aged under 30 Patient can not answer the self-administered questionnaire Patient has not agreed to participate in the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient suffering from Parkinson's disease
Sampling Method: Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Quality of life | 2 years
  Self questionnaires with Beck Depression Scale
Quality of life | 2 years
  use of measurement scales Quality of Life; PDQ-39 it's a 39-item Parkinson's disease questionnaire (Record socio-demographic information)

SECONDARY OUTCOMES:
Socio-demographic data | 2 years
  age, sex, socioeconomic status,
clinical evaluation | 2 years
  clinical form of the disease
clinical evaluation | 2 years
  current treatments and comorbidities
clinical evaluation | 2 years
  Questionnaire administered hetero Q1, Early questionnaire and UPDRS (Unified Parkinson's Disease Rating Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique des Hôpitaux de Marseille